CLINICAL TRIAL: NCT07026292
Title: A Phase Ⅲ, Multicenter, Prospective, Open-Label, Controlled Study of Supermicrosurgical Lymphaticovenous Anastomosis for Prevention of Upper Limb Lymphedema in Breast Cancer Patients Following Axillary Lymph Node Dissection and Adjuvant Radiotherapy
Brief Title: Supermicrosurgical Lymphaticovenous Anastomosis for Prevention of Upper Limb Lymphedema
Acronym: SLVA-PULL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E20250412; TZ3582023-013 (Other Grant/Funding Number: Tianjin Medical University Cancer Institute and Hospital)
Record Dates: First submitted 2025-05-24; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer-Related Lymphedema; Lymphedema; Breast Cancer Invasive
Keywords: Supermicrosurgical Lymphaticovenous Anastomosis; Lymphedema; Breast Cancer; Prevention; Immediate Distal Lymphaticovenous Anastomosis
MeSH Terms: conditions — Breast Cancer Lymphedema; Lymphedema; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ID-LVA Group (Experimental): Immediate distal lymphaticovenous anastomosis (ID-LVA) performed concomitantly with axillary lymph node dissection (ALND)
  Interventions: Procedure: Immediate Distal Lymphaticovenous Anastomosis (ID-LVA)
- non-ID-LVA Group (No Intervention): Axillary lymph node dissection (ALND) without concurrent immediate distal lymphaticovenous anastomosis (ID-LVA)

INTERVENTIONS:
Procedure: Immediate Distal Lymphaticovenous Anastomosis (ID-LVA) — ID-LVA (Immediate Distal Lymphaticovenous Anastomosis) is an supermicrosurgical technique performed during axillary lymph node dissection (ALND) to prevent breast cancer-related lymphedema, offering the dual advantages of immediate intervention and radiation-field avoidance. Compared to LYMPHA (Lymphatic Microsurgical Preventive Healing Approach), which utilizes proximal axillary anastomoses within the radiation field with larger vessels and higher venous pressure, ID-LVA creates precise anastomoses between 0.3-0.8mm distal superficial lymphatic vessels and low-pressure venules in the upper arm. In contrast to DD-LVA (Delayed Distal Lymphaticovenous Anastomosis) performed postoperatively (typically 4-12 weeks after ALND) for subclinical lymphedema, ID-LVA provides earlier prevention by utilizing undamaged lymphatics and avoids the need for a second procedure.
  Other Names: Supermicrosurgical Lymphaticovenous Anastomosis
  Arms: ID-LVA Group

SUMMARY:
Breast cancer-related lymphedema (BCRL) is one of the most common chronic complications following breast cancer treatment. This study enrolls breast cancer patients who are required to undergo axillary lymph node dissection and postoperative adjuvant radiotherapy. Based on patients' preferences, they will be assigned to receive either immediate distal lymphaticovenous anastomosis (ID-LVA) following axillary lymph node dissection (experimental group) or not (control group). The study aims to evaluate the safety and efficacy of ID-LVA in preventing breast cancer-related upper limb lymphedema.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 years;
2. Female;
3. Pathologically confirmed invasive breast cancer;
4. Unilateral breast cancer;
5. Clinical stage T1-4 and N1-3 (post-neoadjuvant therapy staging for patients receiving neoadjuvant treatment);
6. No clinical or radiographic evidence of distant metastasis;
7. Scheduled to undergo axillary lymph node dissection with planned adjuvant radiotherapy;
8. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Currently participating in other clinical trials that, in the investigator's judgment, may affect upper limb lymphatic drainage.
2. No definitive indication for axillary lymph node dissection or adjuvant radiotherapy after neoadjuvant therapy.
3. Pregnant or lactating women.
4. Patients undergoing concurrent autologous tissue flap breast reconstruction or chest wall repair.
5. Upper limb deformities, prior upper limb trauma, or surgical history that, in the investigator's assessment, may compromise lymphatic drainage.
6. Pre-existing upper limb lymphedema at baseline.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Lymphedema incidence | From enrollment to 24 months after surgery
  Breast cancer-related lymphedema (BCRL) was assessed using relative volume change (RVC) derived from circumferential measurements of both upper limbs. Certified lymphedema therapists performed standardized measurements at anatomical landmarks: the web space, ulnar styloid midpoint, and points 10, 20, 30, and 40 cm above the ulnar styloid; axillary measurements were added if needed. Segmental volumes were calculated using the truncated cone formula: V = (πh/12) × (C₁² + C₁C₂ + C₂²), where h = 10 cm, and C₁, C₂ are circumferences at segment ends. Total arm volume was the sum of all segments. RVC was computed as: RVC = (A₂U₁) / (A₁U₂) × 100%, where A₁/A₂ = pre-/postoperative volume of the affected arm, and U₁/U₂ = pre-/postoperative volume of the unaffected arm. If weight fluctuated significantly, weight-adjusted change (WAC) was calculated: WAC = (A₂ × W₁) / (W₂ × A₁) - 1, where W₁ and W₂ represent the preoperative and postoperative body weight.

SECONDARY OUTCOMES:
Lymphedema Severity | From enrollment to 24 months after surgery
  The severity of lymphedema is classified into stages 0 to Ⅲ by breast surgeons and lymphedema therapists according to the International Society of Lymphology (ISL) staging system.
Lymphedema-Associated Symptoms | From enrollment to 24 months after surgery
  Upper limb lymphedema symptoms were assessed using a patient self-reported format. The Breast Cancer and Lymphedema Symptom Experience Index (BCLE-SEI), developed by Fu et al., was employed to evaluate patients' experiences of lymphedema-related symptoms. The scale consists of two components: symptom occurrence and symptom distress. In this study, only the symptom occurrence component was used, which includes 24 items. Each item is rated on a 5-point Likert scale (0 = not at all to 4 = very much), yielding a total score ranging from 0 to 96. Higher scores indicate more severe symptoms. Additionally, each item can be treated as a categorical variable based on the presence or absence of the symptom. The Cronbach's alpha coefficient for this scale is 0.930.
Quality of Life (QoL) | From enrollment to 24 months after surgery
  Quality of life was evaluated using the Functional Assessment of Cancer Therapy - Breast (FACT-B), a validated patient-reported outcome measure developed by David Cella and colleagues as part of the Functional Assessment of Chronic Illness Therapy (FACIT) system, under the Center on Outcomes, Research and Education (CORE) at Northwestern University, United States. The FACT-B consists of 36 items across five domains: physical well-being, social/family well-being, emotional well-being, functional well-being, and additional concerns. Each item is rated on a 4-point Likert scale (0 = not at all to 4 = very much), with higher scores indicating better quality of life. The Chinese version was translated and culturally adapted by Wan Chonghua et al., with reported Cronbach's alpha coefficients ranging from 0.61 to 0.84.
Surgery-Related Complications | From the day of surgery to 1 month after surgery
Radiation-Related Complications | From the day of radiation to 7 days after radiation
Disease-Free Survival (DFS) | From enrollment to 24 months after surgery
Local Recurrence-Free Survival (LRFS) | From enrollment to 24 months after surgery
Overall Survival (OS) | From enrollment to 24 months after surgery

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial, only IPD used in the results publication.
Supporting Information: Study Protocol
Time Frame: From June 1, 2025 to May 31, 2029.